CLINICAL TRIAL: NCT06887075
Title: Systemic Activation of Inflammasomes and Frailty in Older Candidates to Kidney Transplantation
Acronym: INTRA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2022/31
Record Dates: First submitted 2025-01-22; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-01

CONDITIONS: Chronic Kidney Failure; Frailty; Aging; Inflammation
Keywords: Older persons; End-stage kidney disease; Kidney transplantation; Immune aging; Chronic low-grade inflammation; Inflammasomes; Frailty
MeSH Terms: conditions — Kidney Failure, Chronic; Frailty; Inflammation | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Frail Patients (Active Comparator): Frailty will be measured clinically using reference criteria in the general population and validated in Kidney Transplantation (KT), i.e. predictive of post-KT complications: delayed recovery of graft function, graft function, early re-hospitalization, occurrence of post-operative confusion, mortality.
  Fragile patients present at least 3 out of 5 criteria
  Interventions: Biological: Blood sample; Behavioral: Geriatric assessment standardized
- non frail patients (Active Comparator): Patients will be considered non-fragile if they present 0 to 2 criteria
  Interventions: Biological: Blood sample; Behavioral: Geriatric assessment standardized

INTERVENTIONS:
Biological: Blood sample — * Immunophenotyping of peripheral lymphocytes, with a focus on proportions of naïve / central memory / effector memory / TEMRA cells, and markers of activation and senescence
  * Serum inflammatory markers : CRP, IL-6, MCP-1, TNF, sTNFR1
  * Single Molecule Array for IL1 and LUMINEX for IL18 in patient's sera
  * RT-qPCR for inflammasomes genes (NLRP3, NLRC4, NLRC5, AIM2, ASC, casp1, IL1b, IL18) expression among peripheral blood mononuclear cells
  * Assembly of the inflammasome platform will be measured in monocytes using intra-cellular staining of the ASC protein and flow cytometry
Behavioral: Geriatric assessment standardized — * Exhaustion (2 standardized questions)
  * Physical activity <383 kcal/week (men) or <270 kcal/week (women), measured using a standardized questionnaire (IPAQ)
  * 4-meters gait speed, with sex and height-specific cutoffs
  * Handgrip strength, measured using a dynamometer, with sex and BMI-sp Comorbidity (CIRS-G score )
  * Screening for intrinsic capacity decline (first step of ICOPE program, adapted to the study, )
  * Physical performance (SPPB score )
  * Cognitive functions (MoCA score ),
  * Depression (GDS-15 score ),
  * Nutrition (MNA score )
  * Sensory functions (Snellen test for vision, HHIES questionnaire for hearing) -- Dependency in activities of daily living (ADL and IADL scores)

SUMMARY:
Kidney transplantation (KT) benefit-risk ratio assessment is a challenge in a growing population of older patients with end-stage kidney disease. A pre-KT frailty phenotype has been found predictive of post-KT complications, but biological mechanisms of frailty are poorly known is these patients. Frailty is associated with chronic low-grade inflammation in the older general population, possibly through the inflammasome pathway. Our main objective is to assess if systemic activation of inflammasomes is associated with frailty in older candidates to KT.

DETAILED DESCRIPTION:
Kidney transplantation (KT) benefit-risk ratio assessment is a challenge in a growing population of older patients with end-stage kidney disease. Chronic low-grade inflammation is a hallmark of biological aging and is associated with age-related diseases and frailty. Frailty is conceptually defined as an agerelated reduction in physiological reserve increasing vulnerability to stressors. A pre-KT frailty phenotype is associated with post-KT complications, including re-hospitalizations, delayed graft function, delirium and 5-year mortality. Taking pre-KT inflammation into account (serum level of CRP, IL6, sTNFR1) improves prediction of mortality on KT waiting-list, independently of comorbidity.

Molecular and cellular pathways of this inflammation are poorly known, and may involve inflammasomes. Inflammasomes are intra-cellular protein complexes whose assembly, upon stress signals, triggers maturation and release of pro-inflammatory cytokines named interleukine (IL)-1 and IL-18. Inflammasomes are involved in locomotor, cognitive and immune aging in mice, and systemic expression of inflammasomes genes is associated with mortality in older humans. Data is lacking about systemic activation of inflammasomes in older patients with end-stage kidney disease. Our main objective is to assess if pre-KT systemic activation of inflammasomes is associated with frailty in older candidates to KT.

We will measure systemic activation of inflammasomes in peripheral blood of older candidates to KT using cytokine bead-based multiplex assay, Single Molecule Array, intra-cytoplasmic staining, flow cytometry and RT-qPCR in peripheral blood mononuclear cells. Frailty will be measured using validated standardized criteria. A frailty phenotype is defined by at least 3 of the following criteria:

weight loss, exhaustion, muscle weakness, low physical activity, low gait speed.

ELIGIBILITY:
* Inclusion criteria:

  * Age ≥ 70
  * Patient candidate to kidney transplantation (during assessment for inscription on the waiting-list, or during waiting time after effective inscription), without absolute contraindication
  * Free, informed and written consent signed by the participant and the investigator (at the latest, on the day of inclusion and before any examination required by the research).
  * Person affiliated or beneficiary of a social security scheme
* Exclusion criteria:

  * Inclusion in an industrial study refusing co-inclusion in our study
  * Person under guardianship, assisted decision-making or under temporary guardianship

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
IL1 | at recruitment (up to 30 days)
  Single Molecule Array for IL1
IL18 | at recruitment (up to 30 days)
  LUMINEX for IL18 in patient's sera
inflammasomes genes | at recruitment (up to 30 days)
  RT-qPCR for inflammasomes genes (NLRP3, NLRC4, NLRC5, AIM2, ASC, casp1, IL1b, IL18) expression among peripheral blood mononuclear cells
inflammasome platform | at recruitment (up to 30 days)
  Assembly of the inflammasome platform will be measured in monocytes using intra-cellular staining of the ASC protein and flow cytometry
Weight | at enrollment (Day 0), at recruitment (up to 30 days)
  Frailty phenotype : Weight loss (unintentional, >4,5 kg during past year)
Activity | at enrollment (Day 0), at recruitment (up to 30 days)
  Frailty phenotype : Physical activity <383 kcal/week (men) or <270 kcal/week (women), measured using a standardized questionnaire (IPAQ)
Gait | at enrollment (day 0), at recruitment (up to 30 days)
  Frailty phenotype : 4-meters gait speed, with sex and height-specific cutoffs
Handgrip strength | at enrollment (day 0), at recruitment (up to 30 days)
  Frailty phenotype : Handgrip strength, measured using a dynamometer, with sex and BMI-specific cutoffs

SECONDARY OUTCOMES:
Comorbidity | at recruitment (up to 30 days)
  Comorbidity : Cumulative Illness Rating Scale (CIRS-G score)
decline | at recruitment (up to 30 days)
  Screening for intrinsic capacity decline : first step of ICOPE program, adapted to the study
Physical performance | at recruitment (up to 30 days)
  Physical performance : Short Physical Performance Battery (SPPB) score. The SPPB (Short Physical Performance Battery) is the sum of scores on three criteria: the balance test, the walking speed test and the chair lift test. This test assesses an individual's physical performance.
  The sum of the scores for all the tests gives an overall performance score. A score below 8 indicates a risk of sarcopenia (or age-related muscular dystrophy).
Cognitive functions | at recruitment (up to 30 days)
  Cognitive functions : Score Montreal Cognitive Assessment (MoCA) score The Montreal Cognitive Assessement (MoCA) is the most sensitive rapid assessment test, providing the most comprehensive evaluation (attention, concentration, executive functions, memory, language, capacitive-vesuo-constructive, abstraction, calculation, orientation) cognitive functions. It is tending to replace the MMSE in clinical practice.
  A score of 26 (25 if cultural level ≤3 = primary diploma = CEP) is considered abnormal.
Depression | at recruitment (up to 30 days)
  Depression : Geriatric Depression Scale (GDS-15 score) 0 - 5 points: normal 5-10 points: mild to moderate depression 11-15 points: severe depression
Nutrition | at recruitment (up to 30 days)
  Nutrition : Mini Nutritional Assessment (MNA score)
  * 12-14 points: MNA score indicates normal nutritional status.
  * 8-11 points: the MNA score indicates a risk of malnutrition.
  * 0-7 points: MNA score indicates malnutrition.
Snellen test | at recruitment (up to 30 days)
  Sensory functions : Snellen test for vision
ADL | at recruitment (up to 30 days)
  Dependency in activities of daily living : Activities of Daily Living ADL The original ADL scale scores each of the 6 items in 0/1, with 1 corresponding to independence and 0 to dependence. The total score ranges from 0 to 6.
  An overall score can be calculated, ranging from 0 (totally dependent) to 6 (best possible independence).
Immunophenotyping | at recruitment (up to 30 days)
  Immunophenotyping of peripheral lymphocytes, with a focus on proportions of naïve / central memory / effector memory / TEMRA cells, and markers of activation and senescence
CRP | at recruitment (up to 30 days)
  Serum inflammatory markers : CRP
IL-6 | at recruitment (up to 30 days)
  Serum inflammatory markers : IL-6
MCP-1 | at recruitment (up to 30 days)
  Serum inflammatory markers : MCP-1
TNF | at recruitment (up to 30 days)
  Serum inflammatory markers : TNF
sTNFR1 | at recruitment (up to 30 days)
  Serum inflammatory markers : sTNFR1
HHIES questionnaire | at recruitment (up to 30 days)
  Sensory functions : Hearing Handicap Inventory for the Elderly Screening (HHIES) questionnaire for hearing. The higher the score, the greater the likelihood of hearing loss
IADL | at recruitment (up to 30 days)
  Dependency in activities of daily living : IADL scores

CONTACTS AND LOCATIONS:
Overall Officials: Florent GUERVILLE, MD, Principal Investigator — University Hospital, Bordeaux
Locations (3):
- France (3):
  - CHU de Bordeaux - Hôpital Pellegrin -, Bordeaux, France
  - CHU de Bordeaux, Hôpital Xavier Arnozan- Gérontologie Clinique, Pessac, France
  - CHU de Toulouse - Hôpital Rangueil, Toulouse, France